CLINICAL TRIAL: NCT01724346
Title: An Open-label Extension Study in Patients 65 Years or Older With Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL) Who Participated in Study PCYC-1115-CA (Ibrutinib Versus Chlorambucil)
Brief Title: Open-label Extension Study in Patients 65 Years or Older With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1116-CA; 2012-003968-44 (EudraCT Number)
Record Dates: First submitted 2012-11-02; First posted 2012-11-09 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: CLL; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Masking Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chlorambucil (Experimental): Participants who received chlorambucil 0.5 mg/kg (to maximum 0.8 mg/kg) Days 1 and 15 of 28-day cycle up to 12 cycles in Study 1115. In Study 1116, participants had the option to crossover to next-line ibrutinib 420 mg/day after disease progression (PD).
  Interventions: Drug: Ibrutinib
- Ibrutinib (Experimental): Participants who received ibrutinib 420 mg daily in Study 1115 received ibrutinib orally once daily. Participants continuing in first-line ibrutinib therapy entered Study 1116 at the ibrutinib dose tolerated in Study 1115.
  Interventions: Drug: Next-line ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib 420 mg (3 x 140-mg capsules) is administered orally once daily
  Other Names: PCI-32765
  Arms: Chlorambucil
Drug: Next-line ibrutinib — Ibrutinib 420 mg (3 x 140-mg capsules) is administered orally once daily
  Other Names: PCI-32765
  Arms: Ibrutinib

SUMMARY:
An Open-label Extension Study in Patients 65 Years or Older with Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL) Who Participated in Study PCYC-1115-CA (Ibrutinib versus Chlorambucil)

ELIGIBILITY:
Inclusion Criteria:

1. Randomized in the parent study, PCYC-1115-CA
2. Informed consent for Study PCYC-1116-CA
3. Independent review committee (IRC)-confirmed disease progression (PD) in the parent study PCYC-1115-CA or closure of the parent study

Exclusion Criteria:

1. Disease progression involving the central nervous system (CNS) or transformation to another histology
2. Intervening chemotherapy, immunotherapy, or investigational agent specifically to treat CLL if administered before date of IRC confirmed progressive disease
3. In the 4 weeks before dosing: radiation therapy, major surgery, or receipt of an investigational drug
4. Requirement for treatment with a strong CYP3A inhibitor
5. Uncontrolled systemic infection or requirement for IV antibiotics
6. Noncompliance on the parent study(PCYC-1115-CA)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 269 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (88):
- United States (16):
  - City of Hope /ID# 1116-0047, Duarte, California
  - Moores Cancer Center at UC San Diego /ID# 1116-0408, La Jolla, California
  - Stanford University/Stanford Cancer Center, Campus Drive /ID# 1116-0038, Stanford, California
  - University of Chicago /ID# 1116-0126, Chicago, Illinois
  - Norton Cancer Institute - St Matthews /ID# 1116-0071, Louisville, Kentucky
  - Comprehensive Cancer Centers of Nevada /ID# 1116-0712, Henderson, Louisiana
  - University of Massachusetts - Worcester /ID# 1116-0307, Worcester, Massachusetts
  - Washington University-School of Medicine /ID# 1116-0221, St Louis, Missouri
  - Northwell Health/Long Island Jewish Hospital /ID# 1116-0350, New Hyde Park, New York
  - University of Rochester Medical Center /ID# 1116-0127, Rochester, New York
  - Southeastern Medical Oncology Center /ID# 1116-0656, Goldsboro, North Carolina
  - Kaiser Permanente - Northwest /ID# 1116-0677, Portland, Oregon
  - University of Pittsburgh - UPMC (Hillman Cancer Center) /ID# 1116-0050, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center /ID# 1116-0032, Houston, Texas
  - Oncology of San Antonio /ID# 1116-0653, San Antonio, Texas
  - Providence St. Mary Regional Cancer Center /ID# 1116-0731, Walla Walla, Washington
- Australia (8):
  - St George Hospital /ID# 1116-0654, Kogarah, New South Wales
  - Princess Alexandra Hospital /ID# 1116-0503, Woolloongabba, Queensland
  - Flinders Medical Centre /ID# 1116-0163, Bedford Park, South Australia
  - Royal Hobart /ID# 1116-0555, Hobart, Tasmania
  - Box Hill Hospital /ID# 1116-0193, Box Hill, Victoria
  - Monash Medical Centre /ID# 1116-0556, Clayton, Victoria
  - St Vincent's Hospital Melbourne /ID# 1116-0501, Fitzroy Melbourne, Victoria
  - Austin Health /ID# 1116-0170, Heidelberg, Victoria
- Belgium (4):
  - ZNA Cadix /ID# 1116-0561, Antwerp, Antwerpen
  - UCL Saint-Luc /ID# 1116-0164, Woluwe-Saint-Lambert, Brussels Capital
  - UZ Gent /ID# 1116-0560, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 1116-0559, Leuven, Vlaams-Brabant
- Canada (2):
  - Tom Baker Cancer Centre /ID# 1116-0157, Calgary, Alberta
  - Cross Cancer Institute /ID# 1116-0018, Edmonton, Alberta
- China (4):
  - Beijing Cancer Hospital /ID# 1116-0670, Beijing, Beijing Municipality
  - Peking University Third Hospital /ID# 1116-0673, Beijing, Beijing Municipality
  - Jiangsu Province Hospital /ID# 1116-0671, Nanjing, Jiangsu
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 1116-0675, Hangzhou, Zhejiang
- Czechia (3):
  - Fakultni nemocnice Brno /ID# 1116-0562, Brno
  - Fakultni nemocnice Hradec Kralove /ID# 1116-0564, Hradec Králové
  - Fakultni nemocnice Plzen /ID# 1116-0566, Pilsen
- Ireland (2):
  - St James Hospital /ID# 1116-0570, Dublin, Dublin
  - University Hospital Galway /ID# 1116-0571, Galway
- Israel (6):
  - Rambam Health Care Campus /ID# 1116-0576, Haifa, H_efa
  - Bnai Zion Medical Center /ID# 1116-0573, Haifa, H_efa
  - Rabin Medical Center /ID# 1116-0575, Haifa, H_efa
  - Shaare Zedek Medical Center /ID# 1116-0577, Jerusalem, Jerusalem
  - Galilee Medical Center /ID# 1116-0578, Nahariya, Northern District
  - Tel Aviv Sourasky Medical Center /ID# 1116-0856, Tel Aviv
- Italy (9):
  - Institute of Hematology Seràgnoli /ID# 1116-0580, Bologna, Emilia-Romagna
  - Ospedale San Raffaele IRCCS /ID# 1116-0523, Milan, Milano
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 1116-0581, Milan, Milano
  - Università La Sapienza /ID# 1116-0583, Rome, Roma
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 1116-0584, Milan
  - Azienda Ospedaliero-Universitaria di Modena /ID# 1116-0524, Modena
  - Azienda Ospedaliero Universitaria Maggiore della Carita di Novara /ID# 1116-0582, Novara
  - Universita degli Studi di Padova /ID# 1116-0527, Padua
  - Policlinico Universitario A Gemelli /ID# 1116-0891, Rome
- New Zealand (5):
  - Auckland City Hospital /ID# 1116-0588, Grafton, Auckland
  - North Shore Hospital /ID# 1116-0663, Takapuna, Auckland
  - Haematology Waikato Hospital /ID# 1116-0586, Hamilton, Waikato Region
  - Wellington Blood and Cancer Centre /ID# 1116-0587, Wellington South, Wellington Region
  - Canterbury Health Labs Canterbury Disrict Health Board /ID# 1116-0589, Christchurch
- Poland (5):
  - MTZ Clinical Research Sp. z o.o. /ID# 1116-0363, Warsaw, Masovian Voivodeship
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im. ks. B. /ID# 1116-0592, Brzozów, Podkarpackie Voivodeship
  - Samodzielny Publiczny Szpital Klinczny Nr-1- Akademickie Cenrum Klinic /ID# 1116-0529, Gdansk, Pomeranian Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej /ID# 1116-0591, Chorzów, Silesian Voivodeship
  - Medical Univ. of Lodz and Copernicus Memorial Hospital /ID# 1116-0531, Lodz
- State Institution of Health of the Ryazan Regional Clinical Hospital /ID# 1116-0707, Ryazan, Ryazan Oblast, Russia
- Spain (6):
  - Hospital Duran i Reynals /ID# 1116-0604, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 1116-0536, Majadahonda, Madrid
  - Hospital Universitario Vall d'Hebron /ID# 1116-0534, Barcelona
  - Hospital Clinic de Barcelona /ID# 1116-0533, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 1116-0535, Barcelona
  - Hospital Universitario HM Sanchinarro /ID# 1116-0537, Madrid
- Turkey (Türkiye) (5):
  - Gazi Universitesi Tip Fakultes /ID# 1116-0608, Yenimahalle, Ankara
  - Ankara Universitesi Tip Fakultesi Ibn-i Sina /ID# 1116-0606, Ankara
  - Ic Hastaliklari Anabilim Dali/Ege University Medical Faculty /ID# 1116-0714, Izmir
  - Dokuz Eylul University Medical Faculty /ID# 1116-0601, Izmir
  - Erciyes Universiitesi Tip Fakultesi /ID# 1116-0602, Kayseri
- Ukraine (4):
  - CNE Vinnytsya Regional Clinical Hospital named after N.I.Pirogov /ID# 1116-0595, Vinnytsia, Vinnytsia Oblast
  - Communal Nonprofit Enterprise Cherkasy Regional Oncology Dispensary /ID# 1116-0597, Cherkasy
  - Municipal Non-Profit Enterprise City Clinical Hospital 4 of Dnipro City Council /ID# 1116-0594, Dnipro
  - SI Institute of Blood Pathology and Transfusion Medicine of NAMS of Ukraine /ID# 1116-0596, Lviv
- United Kingdom (8):
  - University Hospitals Dorset NHS Foundation Trust /ID# 1116-0551, Poole, Dorset
  - University Hospital Southampton NHS Foundation Trust /ID# 1116-0367, Southampton, Hampshire
  - Nottingham University Hospitals NHS Trust /ID# 1116-0548, Nottingham, Nottinghamshire
  - Oxford University Hospitals NHS Foundation Trust /ID# 1116-0668, Oxford, Oxfordshire
  - Cardiff & Vale University Health Board /ID# 1116-0607, Cardiff, Wales
  - East Suffolk and North Essex NHS Foundation Trust /ID# 1116-0549, Colchester
  - Leeds Teaching Hospitals NHS Trust /ID# 1116-0550, Leeds
  - King's College Hospital NHS Foundation Trust /ID# 1116-0544, London

IPD SHARING:
Plan to Share IPD: Yes
Requests for access to individual participant data from clinical studies conducted by Pharmacyclics LLC, an AbbVie Company, can be submitted through Yale Open Data Access (YODA) Project site at the following link.
URL: http://yoda.yale.edu

REFERENCES:
- [Derived] Burger JA, Barr PM, Robak T, Owen C, Tedeschi A, Sarma A, Patten PEM, Grosicki S, McCarthy H, Offner F, Szafer-Glusman E, Zhou C, Szoke A, Neumayr L, Dean JP, Ghia P, Kipps TJ. Final analysis of the RESONATE-2 study: up to 10 years of follow-up of first-line ibrutinib treatment for CLL/SLL. Blood. 2025 Oct 30;146(18):2168-2176. doi: 10.1182/blood.2024028205. PMID 40737596
- [Derived] Barr PM, Owen C, Robak T, Tedeschi A, Bairey O, Burger JA, Hillmen P, Dearden C, Grosicki S, McCarthy H, Li JY, Offner F, Moreno C, Jermain M, Zhou C, Hsu E, Szoke A, Kipps TJ, Ghia P. Many People With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma Benefit From Ibrutinib Treatment Up To 8 Years: A Plain Language Summary. Future Oncol. 2023 Jan 9. doi: 10.2217/fon-2022-0898. Online ahead of print. PMID 36617990
- [Derived] Barr PM, Owen C, Robak T, Tedeschi A, Bairey O, Burger JA, Hillmen P, Coutre SE, Dearden C, Grosicki S, McCarthy H, Li JY, Offner F, Moreno C, Zhou C, Hsu E, Szoke A, Kipps TJ, Ghia P. Up to 8-year follow-up from RESONATE-2: first-line ibrutinib treatment for patients with chronic lymphocytic leukemia. Blood Adv. 2022 Jun 14;6(11):3440-3450. doi: 10.1182/bloodadvances.2021006434. PMID 35377947
- [Derived] Coutre SE, Byrd JC, Hillmen P, Barrientos JC, Barr PM, Devereux S, Robak T, Kipps TJ, Schuh A, Moreno C, Furman RR, Burger JA, O'Dwyer M, Ghia P, Valentino R, Chang S, Dean JP, James DF, O'Brien SM. Long-term safety of single-agent ibrutinib in patients with chronic lymphocytic leukemia in 3 pivotal studies. Blood Adv. 2019 Jun 25;3(12):1799-1807. doi: 10.1182/bloodadvances.2018028761. PMID 31196847
- [Derived] Barr PM, Robak T, Owen C, Tedeschi A, Bairey O, Bartlett NL, Burger JA, Hillmen P, Coutre S, Devereux S, Grosicki S, McCarthy H, Li J, Simpson D, Offner F, Moreno C, Zhou C, Styles L, James D, Kipps TJ, Ghia P. Sustained efficacy and detailed clinical follow-up of first-line ibrutinib treatment in older patients with chronic lymphocytic leukemia: extended phase 3 results from RESONATE-2. Haematologica. 2018 Sep;103(9):1502-1510. doi: 10.3324/haematol.2018.192328. Epub 2018 Jun 7. PMID 29880603

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This extension study provided ongoing treatment and follow-up for participants previously enrolled in the parent study (PCYC-1115-CA; Study 1115; NCT01722487). Participants entered this study upon Independent Review Committee (IRC)-confirmed progressive disease (PD) or the closure of Study 1115, whichever was earlier.
Pre-assignment Details: All participants randomized to chlorambucil in Study 1115 completed or discontinued their first-line treatment prior to rollover. Participants randomized to ibrutinib in Study 1115 with no PD could continue their first-line treatment in this study. Next-line treatment with ibrutinib after PD was a subsequent-therapy option for participants enrolled in the chlorambucil arm only.
Groups:
- Chlorambucil: Participants who received chlorambucil 0.5 mg/kg (to maximum 0.8 mg/kg) Days 1 and 15 of 28-day cycle up to 12 cycles in Study 1115. In Study 1116, participants had the option to receive next-line ibrutinib 420 mg/day after PD.
Period: Overall Study
Arm/Group | Ibrutinib | Chlorambucil
Started | 136 | 133
Received Next-Line Ibrutinib After PD | 0 (not applicable to this arm) | 78
Completed | 57 | 63
Not Completed | 79 | 70
Not completed — Death | 42 | 42
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 27 | 19
Not completed — Did Not Rollover From Parent Study | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Chlorambucil: Participants who received chlorambucil 0.5 mg/kg (to maximum 0.8 mg/kg) Days 1 and 15 of 28-day cycle up to 12 cycles in Study 1115. In Study 1116, participants had the option to crossover to next-line ibrutinib 420 mg/day after PD.
- Total: Total of all reporting groups
Arm/Group | Ibrutinib | Chlorambucil | Total
Number analyzed (Participants) | 136 | 133 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (5.67) | 73.4 (5.95) | 73.3 (5.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 88 | 81 | 169
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 132 | 129 | 261
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 120 | 125 | 245
  Asian | 9 | 4 | 13
  Black or African American | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Subject declined to answer/unknown | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Based on Investigator Assessment
Description: PFS is defined as the time from the date of randomization to the date of disease progression determined by the investigator or date of death from any cause, whichever occurs first, regardless of the use of subsequent antineoplastic therapy prior to disease progression (PD) or death. Estimated by Kaplan-Meier method.
Time Frame: Median overall follow-up of 82.7 months
Population: Intent-to-Treat (ITT) Population: All randomized participants in Study 1115.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 136 | 133
months | 106.9 [83.4 to NA] — Not estimable because there were not enough PFS events to get a reliable upper bound of 95% confidence interval (CI). | 15.0 [10.2 to 19.4]
Statistical Analysis 1: Comparison: Ibrutinib vs Chlorambucil; Test type: Superiority; p < 0.0001, Log Rank — P-value is from stratified log-rank test; Hazard Ratio (HR) = 0.155, 95% CI 2-sided [0.110 to 0.220]

2. Secondary Outcome: Progression Free Survival After Initiation of Subsequent Anticancer Therapy (PFS2)
Description: PFS2 is defined as the time from the date of randomization to the earliest occurrence of the following three types of events:
  * PD per investigator response assessment after initiation of the first subsequent anti-cancer therapy
  * Initiation of second subsequent anti-cancer therapy
  * Death due to any cause, regardless of administration of subsequent anticancer therapy.
  Kaplan-Meier landmark estimate of the PFS2 rate at 60 months (that is, the estimated percentage of participants with PFS2 at Month 60) is presented.
Time Frame: Median overall follow-up of 82.7 months
Population: ITT Population: All randomized participants in Study 1115.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 136 | 133
percentage of participants | 79.3 [71.1 to 85.4] | 58.4 [48.8 to 66.7]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death due to any cause. Kaplan-Meier landmark estimate of the OS rate at 60 months (that is, the estimated percentage of participants with OS at Month 60) is presented.
Time Frame: Median overall follow-up of 82.7 months
Population: ITT Population: All randomized participants in Study 1115.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 136 | 133
percentage of participants | 82.8 [75.0 to 88.3] | 68.4 [59.1 to 75.9]

4. Secondary Outcome: Time to Next Treatment (TTNT)
Description: Time from randomization to initiation of any subsequent treatment for chronic lymphocytic leukemia (CLL).
Time Frame: Median overall follow-up of 82.7 months
Population: ITT Population: All randomized participants in Study 1115.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 136 | 133
months | NA [NA to NA] — Not estimable because there were not enough TTNT events. | 25.1 [21.8 to 27.9]
Statistical Analysis 1: Comparison: Ibrutinib vs Chlorambucil; Test type: Superiority; p < 0.0001, Log Rank — P value is from stratified log-rank test; Hazard Ratio (HR) = 0.087, 95% CI 2-sided [0.054 to 0.141]

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieve complete response (CR), complete response with an incomplete marrow recovery (CRi), nodular partial response (nPR), or partial response (PR), as determined by the investigator at or prior to initiation of subsequent antineoplastic therapy according to the International Workshop on CLL (iwCLL) 2008 criteria with the 2012 iwCLL modification stating that treatment-related lymphocytosis in the setting of improvement in other parameters was not considered as PD and the 2013 iwCLL clarification of criteria for a partial response to therapy.
Time Frame: Median overall follow-up of 82.7 months
Population: ITT Population: All randomized participants in Study 1115.
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 136 | 133
percentage of participants | 91.2 | 36.8
Statistical Analysis 1: Comparison: Ibrutinib vs Chlorambucil; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Rate ratio and p-value are based on Cochran-Mantel-Haenszel chi-square test stratified by Eastern Cooperative Oncology Group (ECOG; 0-1 vs 2) and Rai stage (0/I/II vs III/IV) at baseline; Rate ratio = 2.496, 95% CI 2-sided [1.990 to 3.131]

6. Secondary Outcome: Rate of Minimal Residual Disease (MRD) Negativity
Description: Percentage of participants who achieved MRD-negative response defined as < 1 CLL cell per 10,000 leukocytes as assessed by flow cytometry of a bone marrow aspirate and/or peripheral blood sample per central laboratory at or prior to initiation of subsequent antineoplastic therapy.
Time Frame: Median overall follow-up of 82.7 months
Population: ITT Population: All randomized participants in Study 1115.
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 136 | 133
percentage of participants | 5.1 | 0

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR will be calculated for the participants achieving a protocol-defined response (Halleck 2008; CR, CRi, nPR, PR) per investigator assessment and is defined as time from the date of initial response including PR with lymphocytosis to the date of disease progression or the date of death from any cause, whichever occurs first.
Time Frame: Median overall follow-up of 82.7 months
Population: ITT Participants Achieving Response (Partial Response or Better) per protocol definitions (Halleck 2008).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib | Chlorambucil
Number analyzed (Participants) | 124 | 49
months | NA [84.0 to NA] — Not estimable because there were not enough DOR events. | 29.7 [15.2 to 40.4]

ADVERSE EVENTS:
Time Frame: All-cause mortality: median overall follow-up of 82.7 months. Adverse events: from first dose of any study treatment to 30 days after last dose of study treatment or initiation of subsequent therapy whichever was earlier. Median treatment duration was: 74.0 months for Ibrutinib arm; 7.1 months for Chlorambucil arm; 26.9 months for Crossover Next-line Ibrutinib arm.
Description: Safety Population: participants in the ITT population who received >= 1 dose of either chlorambucil or ibrutinib as the first-line therapy in the parent Study 1115. The crossover analysis set used for next-line ibrutinib treatment included all chlorambucil arm participants who received at least 1 dose of ibrutinib as the next-line study treatment.
  (Two participants in the Chlorambucil arm died after exiting the study, and are reported here but are not reflected in the Participant Flow table.)
Groups:
- Chlorambucil: Participants who received chlorambucil 0.5 mg/kg (to maximum 0.8 mg/kg) Days 1 and 15 of 28-day cycle up to 12 cycles in Study 1115.
- Next-line Ibrutinib After PD on Chlorambucil: Participants who received chlorambucil treatment in Study 1115 and crossed over to next-line ibrutinib 420 mg/day in Study 1116.
Arm/Group | Ibrutinib | Chlorambucil | Next-line Ibrutinib After PD on Chlorambucil
All-Cause Mortality (participants affected / at risk) | 42/135 | 44/132 | 24/78
Serious Adverse Events (participants affected / at risk) | 111/135 | 33/132 | 49/78
Other Adverse Events (participants affected / at risk) | 134/135 | 120/132 | 75/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib (N=135) | Chlorambucil (N=132) | Next-line Ibrutinib After PD on Chlorambucil (N=78)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 1 (1)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4 (5) | 2 (2) | 2 (2)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (2) | 2 (2) | 2 (2)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
AORTIC VALVE DISEASE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
AORTIC VALVE DISEASE MIXED (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 11 (11) | 1 (1) | 6 (8)
ATRIAL FLUTTER (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 5 (6) | 0 (0) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 (2) | 1 (2) | 0 (0)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
SINUS NODE DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
THYROGLOSSAL CYST (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
BLINDNESS UNILATERAL (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
EYE OEDEMA (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
GLAUCOMA (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
RETINAL VASCULAR OCCLUSION (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
RETINAL VEIN OCCLUSION (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
VITREOUS HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2)
DIVERTICULUM (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
HIATUS HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
MELAENA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OVERFLOW DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 1 (1) | 0 (0)
DEATH (General disorders) | 2 (2) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 3 (3) | 1 (1) | 0 (0)
PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0)
PHYSICAL DECONDITIONING (General disorders) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 4 (6) | 5 (5) | 1 (2)
SUDDEN DEATH (General disorders) | 1 (1) | 0 (0) | 1 (1)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (2) | 0 (0) | 1 (1)
CHOLANGITIS (Hepatobiliary disorders) | 3 (5) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HEPATITIS TOXIC (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 1 (2) | 0 (0) | 0 (0)
IMMUNODEFICIENCY (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ACUTE HEPATITIS B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BACTERIAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BILIARY SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CANDIDA SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 3 (4) | 0 (0) | 2 (2)
CHOLANGITIS INFECTIVE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CHRONIC SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
CORONAVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ESCHERICHIA INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ESCHERICHIA SEPSIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
INFECTED SKIN ULCER (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
KLEBSIELLA INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (5) | 1 (1) | 2 (3)
LOWER RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ORCHITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 27 (38) | 2 (2) | 7 (14)
PNEUMONIA BACTERIAL (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
PNEUMONIA FUNGAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA LEGIONELLA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PULMONARY SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 5 (6) | 0 (0) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 6 (11) | 0 (0) | 5 (5)
UROSEPSIS (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HEAT STROKE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HYPHAEMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SHOULDER FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
FIBRIN D DIMER INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
HEART RATE IRREGULAR (Investigations) | 1 (1) | 0 (0) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 5 (7) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (7) | 0 (0) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMATOMA MUSCLE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (12) | 0 (0) | 1 (1)
BASOSQUAMOUS CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
COLORECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0) | 0 (0)
MUCINOUS ADENOCARCINOMA OF APPENDIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
NON-SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0)
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
RICHTER'S SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
SPINDLE CELL SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (5)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (2)
CAUDA EQUINA SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CEREBELLAR INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2)
COGNITIVE DISORDER (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
DEMENTIA (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
EPILEPSY (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEMIANOPIA HOMONYMOUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
POST HERPETIC NEURALGIA (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 5 (7) | 2 (2) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 5 (6) | 1 (1) | 2 (2)
DEVICE OCCLUSION (Product Issues) | 0 (0) | 0 (0) | 1 (1)
CARDIOVASCULAR SOMATIC SYMPTOM DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
DELIRIUM (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 4 (5) | 0 (0) | 1 (2)
BLADDER CYST (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
BLADDER TAMPONADE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
CALCULUS BLADDER (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (1)
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
RENAL HAEMORRHAGE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
PERINEAL FISTULA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 2 (4) | 2 (2)
PNEUMOMEDIASTINUM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
AORTIC ANEURYSM (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
AORTIC STENOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 4 (4) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib (N=135) | Chlorambucil (N=132) | Next-line Ibrutinib After PD on Chlorambucil (N=78)
ANAEMIA (Blood and lymphatic system disorders) | 33 (86) | 25 (53) | 14 (29)
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 22 (29) | 5 (5) | 8 (8)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 6 (9) | 0 (0) | 4 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 24 (43) | 28 (50) | 7 (17)
SPONTANEOUS HAEMATOMA (Blood and lymphatic system disorders) | 7 (13) | 0 (0) | 4 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 20 (49) | 17 (29) | 8 (9)
ATRIAL FIBRILLATION (Cardiac disorders) | 21 (23) | 0 (0) | 6 (7)
PALPITATIONS (Cardiac disorders) | 11 (13) | 1 (1) | 5 (6)
CATARACT (Eye disorders) | 22 (27) | 2 (2) | 5 (7)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 14 (14) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 27 (40) | 6 (7) | 5 (6)
EYE IRRITATION (Eye disorders) | 13 (23) | 5 (5) | 4 (7)
EYE PAIN (Eye disorders) | 10 (14) | 2 (2) | 3 (4)
LACRIMATION INCREASED (Eye disorders) | 20 (47) | 8 (10) | 6 (10)
PHOTOPHOBIA (Eye disorders) | 8 (10) | 2 (2) | 4 (8)
VISION BLURRED (Eye disorders) | 23 (33) | 11 (11) | 8 (11)
VISUAL ACUITY REDUCED (Eye disorders) | 17 (24) | 3 (3) | 3 (3)
VITREOUS FLOATERS (Eye disorders) | 13 (19) | 7 (8) | 2 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 22 (30) | 13 (13) | 6 (8)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 10 (13) | 6 (7) | 4 (6)
APHTHOUS ULCER (Gastrointestinal disorders) | 7 (7) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 30 (48) | 21 (21) | 12 (14)
DIARRHOEA (Gastrointestinal disorders) | 67 (145) | 22 (33) | 27 (60)
DYSPEPSIA (Gastrointestinal disorders) | 21 (26) | 3 (3) | 11 (11)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 17 (17) | 2 (2) | 3 (3)
HAEMORRHOIDS (Gastrointestinal disorders) | 8 (9) | 3 (3) | 2 (2)
MOUTH ULCERATION (Gastrointestinal disorders) | 9 (9) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 43 (60) | 52 (75) | 13 (22)
STOMATITIS (Gastrointestinal disorders) | 13 (22) | 5 (5) | 2 (3)
VOMITING (Gastrointestinal disorders) | 29 (37) | 27 (42) | 10 (17)
ASTHENIA (General disorders) | 17 (20) | 5 (7) | 9 (12)
CHEST PAIN (General disorders) | 10 (11) | 0 (0) | 4 (6)
FATIGUE (General disorders) | 55 (110) | 51 (85) | 18 (35)
OEDEMA PERIPHERAL (General disorders) | 39 (71) | 11 (11) | 15 (21)
PAIN (General disorders) | 7 (7) | 0 (0) | 3 (4)
PERIPHERAL SWELLING (General disorders) | 7 (10) | 2 (2) | 4 (5)
PYREXIA (General disorders) | 36 (59) | 14 (23) | 9 (20)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 7 (24) | 0 (0) | 3 (11)
BRONCHITIS (Infections and infestations) | 17 (34) | 4 (5) | 5 (7)
COVID-19 (Infections and infestations) | 15 (18) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 13 (17) | 1 (1) | 3 (3)
CONJUNCTIVITIS (Infections and infestations) | 22 (37) | 3 (3) | 8 (11)
CYSTITIS (Infections and infestations) | 7 (11) | 0 (0) | 1 (2)
EYE INFECTION (Infections and infestations) | 8 (9) | 0 (0) | 1 (1)
FOLLICULITIS (Infections and infestations) | 7 (7) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 13 (14) | 7 (8) | 1 (1)
INFLUENZA (Infections and infestations) | 7 (11) | 4 (4) | 7 (9)
NASOPHARYNGITIS (Infections and infestations) | 15 (27) | 6 (6) | 5 (11)
PHARYNGITIS (Infections and infestations) | 8 (9) | 0 (0) | 2 (2)
PNEUMONIA (Infections and infestations) | 12 (16) | 3 (3) | 5 (9)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (8) | 2 (3) | 4 (9)
RHINITIS (Infections and infestations) | 7 (14) | 2 (2) | 0 (0)
SINUSITIS (Infections and infestations) | 9 (14) | 1 (1) | 3 (3)
SKIN INFECTION (Infections and infestations) | 13 (16) | 3 (3) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 38 (73) | 23 (30) | 20 (31)
URINARY TRACT INFECTION (Infections and infestations) | 29 (87) | 10 (15) | 10 (14)
CONTUSION (Injury, poisoning and procedural complications) | 26 (40) | 2 (2) | 4 (4)
FALL (Injury, poisoning and procedural complications) | 25 (45) | 3 (5) | 9 (14)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 8 (8) | 1 (1) | 1 (1)
SKIN ABRASION (Injury, poisoning and procedural complications) | 9 (10) | 1 (1) | 1 (2)
SKIN LACERATION (Injury, poisoning and procedural complications) | 5 (10) | 4 (5) | 4 (4)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 6 (9) | 2 (2) | 4 (5)
BLOOD CREATININE INCREASED (Investigations) | 11 (16) | 2 (3) | 5 (5)
PLATELET COUNT DECREASED (Investigations) | 7 (62) | 6 (10) | 1 (6)
WEIGHT DECREASED (Investigations) | 34 (47) | 16 (16) | 12 (16)
DECREASED APPETITE (Metabolism and nutrition disorders) | 24 (38) | 19 (26) | 7 (10)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 23 (37) | 1 (1) | 2 (5)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 7 (25) | 3 (3) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 16 (26) | 2 (2) | 6 (9)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 7 (15) | 1 (1) | 5 (10)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 12 (14) | 0 (0) | 5 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 41 (75) | 10 (18) | 22 (40)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 27 (38) | 9 (9) | 10 (12)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 7 (9) | 1 (1) | 3 (4)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 28 (40) | 7 (7) | 13 (20)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 9 (10) | 2 (2) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 11 (17) | 4 (6) | 3 (3)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 8 (11) | 4 (5) | 2 (3)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 8 (8) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 23 (27) | 7 (7) | 8 (10)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (22) | 2 (3) | 5 (6)
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (10) | 2 (2) | 1 (1)
DIZZINESS (Nervous system disorders) | 25 (29) | 16 (22) | 10 (14)
HEADACHE (Nervous system disorders) | 19 (32) | 13 (23) | 9 (17)
HYPOAESTHESIA (Nervous system disorders) | 7 (10) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 7 (8) | 1 (1) | 4 (6)
SYNCOPE (Nervous system disorders) | 7 (7) | 2 (2) | 2 (4)
ANXIETY (Psychiatric disorders) | 16 (21) | 2 (2) | 4 (5)
DEPRESSION (Psychiatric disorders) | 11 (11) | 5 (5) | 7 (10)
INSOMNIA (Psychiatric disorders) | 18 (22) | 9 (11) | 6 (11)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 9 (13) | 0 (0) | 2 (2)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 8 (12) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 13 (14) | 3 (3) | 6 (8)
POLLAKIURIA (Renal and urinary disorders) | 8 (8) | 4 (4) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 52 (79) | 20 (24) | 19 (25)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 21 (37) | 13 (16) | 11 (20)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (7) | 4 (4)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 21 (26) | 5 (8) | 7 (8)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 2 (2) | 3 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 16 (23) | 5 (5) | 3 (3)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 11 (17) | 1 (1) | 4 (5)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2) | 3 (3)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 12 (19) | 2 (2) | 2 (2)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 5 (8)
DRY SKIN (Skin and subcutaneous tissue disorders) | 12 (13) | 3 (3) | 4 (7)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1) | 9 (12)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 14 (16) | 10 (12) | 3 (3)
PETECHIAE (Skin and subcutaneous tissue disorders) | 7 (8) | 1 (1) | 5 (5)
PRURITUS (Skin and subcutaneous tissue disorders) | 19 (29) | 7 (13) | 5 (10)
PURPURA (Skin and subcutaneous tissue disorders) | 7 (8) | 0 (0) | 2 (3)
RASH (Skin and subcutaneous tissue disorders) | 9 (22) | 3 (8) | 3 (3)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 17 (30) | 6 (6) | 4 (4)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 13 (19) | 5 (7) | 6 (17)
SKIN LESION (Skin and subcutaneous tissue disorders) | 11 (13) | 1 (1) | 4 (5)
HYPERTENSION (Vascular disorders) | 37 (64) | 0 (0) | 10 (26)
HYPOTENSION (Vascular disorders) | 6 (6) | 6 (8) | 4 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT01724346/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT01724346/SAP_001.pdf